CLINICAL TRIAL: NCT06216392
Title: A Randomized, Double-Blind, Placebo-Controlled, Multi-Center, Phase 3 Trial Evaluating the Efficacy, Safety, and Immunogenicity of GR1802 Injection in Patients With Moderate to Severe Atopic Dermatitis
Brief Title: Phase III Study of GR1802 Injection in Patients With Atopic Dermatitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Genrix (Shanghai) Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GR1802-004
Record Dates: First submitted 2024-01-11; First posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2023-12

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: GR1802 (Experimental): GR1802 injection 300mg every two weeks for 52-week treatment.
  Interventions: Biological: GR1802 injection
- Placebo (Placebo Comparator): Placebo every two weeks for 16-week treatment. Crossover to GR1802 injection for another 36 weeks
  Interventions: Biological: placebo

INTERVENTIONS:
Biological: GR1802 injection — 150mg/1ml. 2 ml every two weeks Route of administration: Subcutaneous
  Arms: Experimental: GR1802
Biological: placebo — 0mg/1ml. 2 ml every two weeks Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double blind, placebo-controlled study to evaluate the efficacy, safety, PK, PD and immumogenicity of GR1802 injection in comparison to placebo in patients with atopic dermatitis. Patients will receive GR1802 injection or Placebo every 2 Weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with AD according to Williams criteria with a history of at least 12 months before Screening, with below requirements: 1) EASI score ≥16 at Screening and Baseline; 2) IGA score ≥3 at Screening and Baseline; 3) ≥10% BSA of AD involvement at Screening and Baseline; 4) Pruritus NRS average score ≥4 at Baseline.
2. Inadequate response or intolerance to topical glucocorticoid therapy for AD within 6 months prior to screening.

Exclusion Criteria:

1. Not enough washing-out period for previous therapy.
2. Concurrent disease/status which may potentially affect the efficacy/safety judgement.
3. Abnormal laboratory test results at screening that, in the judgment of the investigator, may affect the subject's ability to complete the trial.
4. Women who are pregnant or breastfeeding, or planning to become pregnant, breastfeeding during the study.
5. Other

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving EASI-75 at week 16 | at Week 16
  The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe).
Proportion of subjects with IGA score of 0 or 1 and a reduction of IGA score by ≥2 points from baseline at week 16 | at Week 16
  IGA is an assessment instrument used in clinical studies to rate the severity of AD globally, based on a 5-point scale ranging from 0 (clear) to 4 (severe).

SECONDARY OUTCOMES:
Percent change of EASI score from baseline | Baseline up to Week 52
  The EASI is a composite index with scores ranging from 0 to 72. Four AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation], and lichenification) will each be assessed for severity by the investigator on a scale of "0" (absent) through "3" (severe).
Percent change of NRS score from baseline | Baseline up to Week 52
  The range of Pruritus Numerical Rating Scale (NRS) is from 0 (no itch)-10 (worst imaginable itch)
Body surface area (BSA) of involvement of atopic dermatitis | Baseline up to Week 52
  Change from baseline in percent of BSA
Changes from baseline in Dermatology Life Quality Index (DLQI) | Baseline up to Week 52
  The DLQI is a 10-item, validated questionnaire used in clinical practice and clinical trials to assess the impact of AD disease symptoms and treatment on quality of life. It is a 10-question questionnaire with a score of 0 (not at all) to 3 (very much) for each question. A high score is indicative of a poor quality of life.
Incidence of adverse events (AEs), abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing. | Baseline up to Week 60
  Incidence of adverse events (AEs), abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Immunogenicity: anti-drug antibody (ADA) and neutralizing antibody (Nab) | Baseline up to Week 60
  anti-drug antibody (ADA) and neutralizing antibody (Nab)
Changes from baseline in Scoring Atopic Dermatitis Index (SCORAD) | Baseline up to Week 52
  SCORAD ("SCORing Atopic Dermatitis") is a clinical tool for assessing the severity (i.e., extent, intensity) of atopic dermatitis as objectively as possible.
Changes from baseline in The Patient-Oriented Eczema Measures for Eczema(POEM) | Baseline up to Week 52
  The Patient Oriented Eczema Measure (POEM) is a tool used for monitoring atopic eczema severity. It focuses on the illness as experienced by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No